CLINICAL TRIAL: NCT01233440
Title: An Open-label, Multicenter, Dose-Escalation Safety and Pharmacokinetic Study of a Recombinant Coagulation Factor IX Albumin Fusion Protein (rIX-FP) in Subjects With Hemophilia B
Brief Title: Safety and Pharmacokinetic Study of a Recombinant Coagulation Factor IX Albumin Fusion Protein in Subjects With Hemophilia B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSL654_2001; 1508 (Other: CSL Behring); 2010-018477-38 (EudraCT Number)
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): 25 IU/kg dose
  Interventions: Biological: Recombinant Coagulation Factor IX Albumin Fusion Protein
- Cohort 2 (Experimental): 50 IU/kg dose
  Interventions: Biological: Recombinant Coagulation Factor IX Albumin Fusion Protein; Biological: Plasma derived FIX [pdFIX]
- Cohort 3 (Experimental): 75 IU/kg dose
  Interventions: Biological: Recombinant Coagulation Factor IX Albumin Fusion Protein

INTERVENTIONS:
Biological: Recombinant Coagulation Factor IX Albumin Fusion Protein — Single dose of 25, 50 or 75 IU/kg of rIX-FP, given as intravenous infusion
Biological: Plasma derived FIX [pdFIX] — Single dose of 50 IU/kg of reference product, given as intravenous infusion
  Arms: Cohort 2

SUMMARY:
The primary objective of the study is to assess the safety of IV administration of rIX-FP. Safety will be evaluated by adverse events and laboratory changes over time. The secondary objective of the study is to evaluate the pharmacokinetics parameters, following a single intravenous dose of rIX-FP.

DETAILED DESCRIPTION:
This study is comprised of both a rIX-FP dose-escalation safety segment (25, 50 and 75 IU/kg of rIX-FP), and PK evaluation of rIX-FP after a single dose of 50 IU/kg, as well as PK evaluation after a single dose of 50 IU/kg of the previously given Factor IX (FIX) product (recombinant FIX [rFIX] or plasma derived FIX [pdFIX]) which is used as the reference product.

ELIGIBILITY:
Inclusion Criteria:

* Male, 12 - 65 years, with body weight ≥ 30 kg and ≤ 120 kg
* Documented severe Hemophilia B (FIX activity of ≤ 2%) or tested by the central laboratory at screening
* Subjects who have received FIX products for > 150 exposure days (EDs) (estimated)
* No confirmed prior history of FIX inhibitor (history of positive FIX inhibitor defined as two consecutive positive tests - a confirmatory test on a second, separately drawn sample shortly after the previous positive test) and confirmed no detectable FIX inhibitors (negative FIX inhibitor defined as < 0.6 Bethesda Units [BU] by the central laboratory at screening
* Subjects can be treated on-demand or under prophylactic therapy
* Signed Informed Consent/Assent

Exclusion Criteria:

* Known hypersensitivity (allergic reaction or anaphylaxis) to any FIX product or hamster protein
* Any known congenital or acquired coagulation disorder other than congenital FIX deficiency
* Platelet count < 100,000/µL
* Immunocompromised (CD4 count < 200/mm3), (HIV positive subjects may participate in the study and protease inhibitors and antiviral therapy are permitted, at the discretion of the Investigator)
* Currently receiving IV immunomodulating agents such as immunoglobulin or chronic systemic corticosteroid treatment
* Serum aspartate aminotransferase (AST) or serum alanine aminotransferase (ALT) concentration > 5 times (x) the upper limit of normal (ULN)
* Serum creatinine > 2 x ULN
* Evidence of thrombosis, including deep vein thrombosis, stroke, pulmonary embolism, myocardial infarction and arterial embolus within 3 months prior to enrollment
* Use of an Investigational Medicinal Product (IMP) within 30 days prior to the first rIX-FP administration
* Experienced life-threatening bleeding episode or had major surgery or an orthopedic surgical procedure during the 3 months prior to study entry
* Subject currently on a dose and/or regimen of FIX that would preclude participation in the study due to possible increased risk of bleeding because of the requirement to withhold treatment during the PK sampling period
* Suspected inability (e.g., language problem or mental condition) or unwillingness to comply with study procedures or history of noncompliance

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) | up to 14 days after drug administration
Frequency of serious adverse events (SAEs) | up to 28 days after drug administration
Occurrence of inhibitor against FIX | up to 28 days after drug administration
Occurrence of antibodies against rIX-FP | up to 28 days after drug administration

SECONDARY OUTCOMES:
AUC to the last sample with quantifiable drug concentration (AUC0-t) | From time of dosing up to 7 days after the dose
  Following 50 IU/kg rIX-FP infusion
AUC extrapolated to infinity (AUCt-∞) | From time of dosing up to 7 days after the dose
  Following 50 IU/kg rIX-FP infusion
Half-life (t1/2) | From time of dosing up to 7 days after the dose
  Following 50 IU/kg rIX-FP infusion
Incremental recovery (IU/mL/IU/kg) | From time of dosing up to 7 days after the dose
  Defined as FIX activity (IU/mL) obtained 30 minutes following infusion, per dose of (IU/kg) infusion.
Clearance | From time of dosing up to 7 days after the dose
  Following 50 IU/kg rIX-FP infusion

CONTACTS AND LOCATIONS:
Overall Officials: Iris Jacobs, MD, Study Director — CSL Behring
Locations (20):
- Study site, Vienna, Austria
- France (4):
  - Study site, Le Kremlin-Bicêtre
  - Study Site, Lyon
  - Study site, Nantes
  - Study site, Paris
- Germany (4):
  - Study Site, Berlin
  - Study Site, Hamburg
  - Study Site, Hanover
  - Study site, Münster
- Study Site, Tel Litwinsky, Israel
- Italy (7):
  - Study Site, Catania
  - Study Site, Florence
  - Study Site, Genova
  - Study site, Milan
  - Study Site, Napoli
  - Study Site, Parma
  - Study Site, Vicenza
- Spain (3):
  - Study Site, A Coruña
  - Study Site, Barcelona
  - Study Site, Madrid

REFERENCES:
- [Derived] Santagostino E, Negrier C, Klamroth R, Tiede A, Pabinger-Fasching I, Voigt C, Jacobs I, Morfini M. Safety and pharmacokinetics of a novel recombinant fusion protein linking coagulation factor IX with albumin (rIX-FP) in hemophilia B patients. Blood. 2012 Sep 20;120(12):2405-11. doi: 10.1182/blood-2012-05-429688. Epub 2012 Aug 2. PMID 22859609